CLINICAL TRIAL: NCT04277702
Title: The Assessment of Cysteinyl Leukotriene Receptor Antagonist Role in Inhibition of Atherosclerosis, Proliferation and Its Influence on Endothelial Function in Patients Undergoing Endovascular Treatment Due to Peripheral Arterial Disease.
Brief Title: Cysteinyl Leukotriene Antagonist in Atherosclerosis Inhibition in Patients After Endovascular Treatment Due to Peripheral Arterial Disease
Acronym: CADET-PAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Pawel Maga, Prof., Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CADET-PAD; 2020-000715-71 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Lower Limb Ischemia; Atherosclerosis of Artery
Keywords: atherosclerosis; Peripheral Arterial Disease; Montelukast; Leukotrienes
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Atherosclerosis | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast + standard treatment (Experimental)
  Interventions: Drug: Montelukast 10mg; Procedure: Endovascular treatment; Drug: Standard anti-platelet treatment
- Placebo+ standard treatment (Placebo Comparator)
  Interventions: Procedure: Endovascular treatment; Drug: Standard anti-platelet treatment

INTERVENTIONS:
Drug: Montelukast 10mg — Oral administration of 10mg of montelukast daily for 12 months
  Arms: Montelukast + standard treatment
Procedure: Endovascular treatment — Percutaneous transluminal angioplasty combined with bare-metal stenting of lower limbs arteries
Drug: Standard anti-platelet treatment — Standard antithrombotic treatment for patients undergoing endovascular procedures

SUMMARY:
Atherosclerosis is a civilization disease, which pathophysiology is based on chronic inflammatory response in the wall of vessels that is caused by increase of pro-inflammatory substances. It is a significant challenge for diagnostics and pharmacology. This disease occurs in over 60% of the population over 70 years old. There are many factors that are responsible for this process including group of the arachidonic acid metabolism products - leukotriens, especially leukotriene E4 (LTE4). The effect of these factors was described as the base of pathology not only cardiovascular diseases but also the base of development of asthma and other allergic diseases. The substance which blocks the activity of these factors - montelukast - is a common method of treatment in asthma.

The aim of this project is to investigate the influence of cysteinyl leukotriens receptor antagonists on lower limb arteries reocclusion rate in patients with peripheral artery disease (PAD) after endovascular treatment.

During previous years we conducted a prospective study, which helped us evaluating the dynamics of leukotriens and thromboxane levels in patients with PAD, who underwent endovascular treatment - peripheral transluminal angioplasty (PTA). We established for the first time the dependence between the increased level of LTE4 in urine (uLTE4) and restenosis or reocclusion occurrence, which translates to the necessity of further procedures and a decrease in the quality of life. We should ask ourselves a question: Is blocking of cysteinyl leukotriens reaction as proinflammatory and proliferative factors, by the use of receptor CysLT1 antagonists going to decrease the quantity of restenosis and reocclusions after endovascular treatment? Within the project performed in the Angiology Department of Jagiellonian University among the patients suffering from PAD and fulfilling all inclusion criteria, the randomized double-blinded clinical study will be performed. Patients will be assigned to two groups: Treatment Group (which will be receiving cysteinyl leukotriene antagonist (montelukast) in a dose of 10mg/day for 12 months) and Control Group to which placebo will be administered. Among all patients population, at every visit at 1., 3., 6., and 12-month clinical state, ultrasound, hemodynamic parameters, and endothelium imaging will be performed as well as uLTE4 measurements. A comparison of the results between both groups will give us an answer if blocking uLTE4 receptors may become a breakthrough in future atherosclerosis treatment.

The mechanisms, which lead to restenosis is still not fully understood, and currently used methods of treatment - antiplatelets, anti-proliferative drugs, and anticoagulants - are not fully effective. Thanks to this research the knowledge about treatment and prevention of atherosclerosis will be increased, which will be connected with future better patient care, especially patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with peripheral arterial disease qualified for endovascular treatment with Rutherford 3 or 4 clinical symptoms.
2. Age 45 - 75 years old.
3. Signed informed consent.

Exclusion Criteria:

1. Patients with peripheral arterial disease (PAOD) with Rutherford 1,2,5 or 6 clinical symptoms.
2. Age < 45 or > 75 years old.
3. Infection and/or fever (temperature above 37,2 C) within the last 3 weeks preceding the study recruitment (viral infections, cold, sinusitis) and use of antibiotics within the last 2 months.
4. Symptoms of acute tissue infection
5. Chronic inflammatory disease (e.g. COPD stage >II in GOLD classification)
6. HIV+, HCV+, HBS+.
7. Autoimmunological diseases and use of steroids or immunosuppressive medications within the last 3 months.
8. Inflammatory blood vessel disorders (with exception of atherosclerosis)
9. Myocardial infarction or stoke within last 6 months.
10. Buerger Disease.
11. Chronic heart failure (3-4 NYHA)
12. Acute lower limb ischemia or surgical revascularization within last 6 months.
13. Serious trauma or surgery procedure within last 6 months.
14. Asthma.
15. On-going antileukotriene treatment.
16. Neoplasm diagnosed within 5 years.
17. Chronic Kidney Disease (creat. >177 µmol/l).
18. Pregnancy, puerperium, women without efficient contraception.
19. Vaccinations within 30 days before recruitment.
20. Hospitalisation in intensive care unit within 3 months.
21. Lack of the possibility of the follow-up participation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Failure of endovascular treatment (Target Vessel Failure) | 12 months
  Hemodynamically significant restenosis or reocclusion of the treated vessel

SECONDARY OUTCOMES:
Death | 12 months
Myocardial Infarction | 12 months
Stroke | 12 months
Combined MACEs | 12 months
  Occurrence of any major adverse cardiovascular event
Treated limb amputation | 12 months
  Large amputation of the treated limb
Significant decrease of life quality | 12 months
  Significant decrease of life quality in patients undergoing treatment measured by the Vascu-Qol and Walking Impairment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Maga, Prof, Principal Investigator — Angiology Department, Jagiellonian University Medical College

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol